CLINICAL TRIAL: NCT01500096
Title: American Ginseng to Improve HIV-Associated Fatigue: A Randomized, Placebo-Controlled, Multiple-Dose Escalation Clinical Trial
Brief Title: American Ginseng to Improve HIV-Associated Fatigue: A Randomized, Placebo-Controlled, Parallel Design, Multiple-Dose Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00071671
Record Dates: First submitted 2011-12-14; First posted 2011-12-26 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: HIV/AIDS-associated Fatigue
Keywords: Fatigue; HIV/AIDS; American ginseng; Panax quinquefolius; Fatigue Severity Scale; CD4 count; plasma HIV RNA; cytokines; IL-6; sTNFR1; sTNFR2
MeSH Terms: conditions — Fatigue; Acquired Immunodeficiency Syndrome | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- American ginseng 1000 mg/day (Active Comparator): 4-week of American ginseng 1000 mg/day every morning
  Interventions: Drug: American ginseng
- Placebo for American ginseng 1000 mg/day (Placebo Comparator): 4-week of placebo for American ginseng 1000 mg/day every morning
  Interventions: Dietary Supplement: Placebo for American ginseng
- American ginseng 3000 mg/day (Active Comparator): 4-week of American ginseng 3000 mg/day every morning
  Interventions: Drug: American ginseng
- Placebo for American ginseng 3000 mg/day (Placebo Comparator): 4-week of placebo for American ginseng 3000 mg/day every morning
  Interventions: Dietary Supplement: Placebo for American ginseng

INTERVENTIONS:
Drug: American ginseng — American ginseng 1000 mg/day and 3000 mg/day will be evaluated in the intervention arms for this study. Participants will be randomized to American ginseng 1000 or 3000 mg/day capsules taken daily for four weeks.
  Other Names: Panax quinquefolius
  Arms: American ginseng 1000 mg/day; American ginseng 3000 mg/day
Dietary Supplement: Placebo for American ginseng — Placebo for American ginseng 1000 mg/day and 3000 mg/day will be evaluated in the control arms for this study. Participants will be randomized to placebo for American ginseng 1000 or 3000 mg/day capsules taken daily for four weeks.
  Arms: Placebo for American ginseng 1000 mg/day, Placebo for American ginseng 3000 mg/day
  Arms: Placebo for American ginseng 1000 mg/day; Placebo for American ginseng 3000 mg/day

SUMMARY:
The purpose of this study is to determine whether American ginseng is effective in the treatment of HIV-associated fatigue.

DETAILED DESCRIPTION:
STUDY DESIGN Chronic fatigue is a major problem for HIV-infected patients and contributes to decreased quality of life and physical functioning, higher levels of psychological distress, and antiretroviral non-adherence. The etiology of fatigue in HIV-infected patients is unknown, but changes in systemic inflammation may play a contributing role. The mechanism of action of ginseng in the treatment of fatigue is also not clear, but in its role as a purported "adaptogen," it may decrease fatigue by altering systemic inflammation. Ginseng is one of the most popular botanical products in the US and is marketed to improve fatigue and vitality. Our preliminary data suggested that American ginseng at 1000-2000 mg/day may decrease fatigue in cancer patients. HIV-infected patients frequently use ginseng, in part because they perceive these therapies to be safer than more conventional therapies.

We hypothesized that a standardized American ginseng formulation will improved HIV-related fatigue. To test this hypothesis we propose a 6-week double-blind, placebo-controlled trial, parallel study of four weeks of treatment involving two doses of American ginseng or placebo (1000mg/day or 3000 mg/day) in 120 HIV-infected patients with clinically significant fatigue, as defined by their scores on the Fatigue Severity Scale. Patients will be treated with American ginseng or placebo every morning for a total of two doses of 1000 mg/day or 3000 mg/day. A smaller cohort of 12 out of 120 subjects will be enrolled initially to monitor closely for confirmed virologic failure, If confirmed virologic failure is not observed, enrollment will continue to the proposed 120 subjects. Virologic failure is defined as two consecutive plasma viral loads >200 cells according to the 2012 Department of Health Humans Services Guidelines for the use of antiretroviral agents in HIV-1 infected adults and adolescents

The proposed doses of American ginseng are the same as those used in our previous trials. American ginseng 1000 mg/day showed efficacy in ameliorating fatigue in cancer patients. The highest dose of American ginseng (3000 mg/day) selected for this study was derived from our previous American ginseng trial.

Change on scores of the Fatigue Severity Scale (FSS) between American ginseng and placebo groups at baseline, and treatment weeks 2, 4, and 6 (the last safety visit two weeks after completing the 4-week treatment period with American ginseng or placebo) will be calculated. The primary comparison of interest will involve the primary endpoint of the average change in the FSS scale score from baseline to the end of treatment. Other instruments to supplement the FSS and further assess fatigue will be a modified version of the Brief Fatigue Inventory (BFI), The Epworth Sleepiness Scale (ESS), the Patient Health Questionnaire (PHQ-9), Insomnia Severity Index (ISI), the Medical Outcomes Study HIV Health Survey (MOS-HIV), the Clinical Global Impressions (CGI) of Change Scale, and Patient-Reported Outcomes Measurement Information System (PROMIS) fatigue. To further elucidate the mechanism of HIV-related fatigue, we will evaluate the effects of American ginseng and placebo on markers of systemic inflammation such as IL-6 and soluble receptors of tumor necrosis factor (TNF) α 1 and 2 (sTNFR1 and sTNFR2), at baseline and weeks 2, 4, and 6. cluster of differentiation 4 (CD4) cell counts, plasma HIV RNA levels, and adverse events (AEs) will also be assessed for safety purposes.

DURATION:

The total duration of this study is 6 weeks. Participants will receive American ginseng or placebo during the first 4 weeks of the study. On week 6 participants will complete their final post treatment safety study visit.

POPULATION AND SAMPLE SIZE:

120 HIV-infected subjects (40 in the American ginseng 1000 mg/day arm, 40 in the American ginseng 3000 mg/day arm, 20 in the placebo 1000 mg/day arm, and 20 in the placebo 3000 mg/day arm).

REGIMEN:

This is a randomized, placebo-controlled, longitudinal, parallel study with two doses of American ginseng. As shown in the study schematic figure, two doses of American ginseng or placebo (1000 or 3000 mg/day) will be given to 120 HIV-infected patients (40 in the American ginseng 1000 mg/day arm, 40 in the American ginseng 3000 mg/day arm, 20 in the placebo 1000 mg/day arm, and 20 in the placebo 3000 mg/day arm) with clinically significant fatigue. Participants will receive American ginseng or placebo for a total of 4 weeks and will be followed for a total of 6 weeks (week 6 is the last safety visit 2 weeks after completing the 4-week treatment period with American ginseng or placebo).

American ginseng will be continued for Grades 1 and 2 toxicities at the discretion of the investigator. Treatment will be discontinued for subjects experiencing any grade ≥3 study drug toxicity. Evaluations for the early termination visit will be completed for these subjects. Participants who discontinue treatment secondary to toxicity will be followed until resolution, return to baseline values, or an adequate explanation can be given for their condition. Subjects requiring dose modifications/reductions/interruptions of American ginseng/placebo to manage toxicities will be followed off study drugs. The total number of patients accrued hence will be 120 patients (40 in the American ginseng 1000 mg/day arm, 40 in the American ginseng 3000 mg/day arm, 20 in the placebo 1000 mg/day arm, and 20 in the placebo American ginseng 3000 mg/day arm).

STUDY DURATION The total duration of this study is six weeks. Participants will receive American ginseng or placebo during the first 4 weeks of the study. On week 6 participants will complete their final post treatment safety study visit.

STUDY AGENT/INTERVENTION DESCRIPTION Two doses of American ginseng or placebo (1000 mg/day or 3000 mg/day) every morning by mouth for a 4-week period.

PRIMARY AND SECONDARY OBJECTIVES The overall objective of this study is to determine the effect of American ginseng on fatigue in HIV-infected subjects. HIV-infected subjects with fatigue will be randomized to receive two doses (1000 mg/day or 3000 mg/day) of standardized American ginseng or placebo, and their levels of fatigue and quality of life will be assessed. We will also quantify proinflammatory cytokines in the placebo and American ginseng-treated groups to further elucidate the mechanism of HIV-related fatigue, and the effects of American ginseng on these markers.

ENDPOINTS

Primary Endpoint: Change in FSS total score from baseline to end of four weeks of treatment.

Secondary Endpoints: Change from baseline and values observed at 2, 4, and 6 weeks post-baseline for the following measures: BFI-global assessment score ESS score PHQ-9 total score ISI score MOS-HIV scale total score, Gene Importance Calculator (GIC) score PROMIS fatigue scale score Serum cytokines (IL-6, sTNFR1, sTNFR2) CD4 cell counts, proportion with detectable plasma HIV RNA, AEs will be measured using the Division of AIDS Table for Grading the Severity of Adults Adverse events.

ELIGIBILITY:
INCLUSION CRITERIA

1. HIV-infected men and women, ≥18 years of age
2. HIV-1 infection documented by a rapid HIV test or any licensed ELISA test kit and confirmed by a repeat ELISA, Western blot at any time prior to study entry; or documentation of ongoing HIV/AIDS care, or treatment for AIDS, or previous positive HIV serology at any time prior to study entry
3. On stable antiretroviral therapy for at least three months
4. Undetectable plasma HIV RNA using conventional assays with lower limits of quantification (20-75 copies/ml) obtained within 30 days prior to entry
5. The following laboratory values obtained within 30 prior to study entry:

   Absolute neutrophil count (ANC) ≥750/mm3 Hematocrit ≥30 Platelet count ≥40,000/mm3 Calculated creatinine clearance (CrCl) ≥50 mL/min, as estimated by the Cockcroft-Gault equation* aspartate amino transferase (AST) serum glutamic oxalacetic transaminase (SGOT), amino alanine transferase (ALT) serum glutamic-pyruvic transaminase (SGPT), and alkaline phosphatase <3 x upper limit of normal (ULN) total bilirubin ≤2.5 x ULN

   NOTE: If the potential subject is taking an atazanavir-containing regimen at the time of screening, total bilirubin ≤5 x ULN is acceptable

   * Calculation for the Cockcroft-Gault equation is available at https://www.fstrf.org/common/utilities/calculators/ccc.html
6. Clinically significant fatigue (≥4.5 on the FSS)
7. PHQ-9 Questionnaire score <10
8. ISI Questionnaire <14
9. On stable psychiatric medications for at least 8 weeks prior to enrollment.
10. Ability and willingness of subject to provide a signed informed consent and comply with all study requirements
11. Laboratory values and physical examination as judged by the principal investigator to be safe to participate
12. Females of reproductive potential (women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy, or bilateral oophorectomy or tubal ligation) will need a negative serum or urine pregnancy test within 30 days prior to entry.

    NOTE: Acceptable documentation of hysterectomy and bilateral oophorectomy, tubal ligation, tubal micro-inserts, and menopause is self-reported history.
13. All potential subjects must agree not to participate in the conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the subject/ partner must reliable methods of contraception (condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an intrauterine contraceptive device (IUD); or hormone-based contraceptive) while receiving study treatment. Subjects will be encourage to use a barrier method of contraception (e.g. condoms) along with hormonal contraceptives during administration of American ginseng.

EXCLUSION CRITERIA

1. Untreated hypothyroidism (TSH >4.5 milli-international units per liter (mIU/L))
2. Untreated or undertreated hypogonadism (calculated free testosterone below The lower limit of normal)
3. Untreated or under-treated major depressive disorder
4. No change in testosterone therapy within 6 weeks prior to screening
5. As determined by the investigator, history of chronic or acute medical condition that in the opinion of the investigator would jeopardize safety of subjects participating in this study
6. Hospitalization or therapy for serious illness within 30 days prior to study entry as judged by the investigator
7. Known allergy/sensitivity or any hypersensitivity to components of American ginseng
8. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence or subject compliance with study requirements (stable methadone treatment allowed)
9. Current use or requirement for any medications prohibited with study treatment including warfarin. (Lists of prohibited medications are contained in the Prohibited Medications Section of the protocol)
10. Pregnancy or breastfeeding
11. Use of any immunomodulator (e.g., interferons, interleukins, systemic corticosteroids, cyclosporine), vaccine, or investigational therapy within 30 days prior to study entry
12. Treatment with investigational study drugs/vaccines
13. Co-enrolment in observational trials is allowed if the blood volume requirement does not exceed the Red Cross limits specified for this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Andrade AS, Hendrix C, Parsons TL, Caballero B, Yuan CS, Flexner CW, Dobs AS, Brown TT. Pharmacokinetic and metabolic effects of American ginseng (Panax quinquefolius) in healthy volunteers receiving the HIV protease inhibitor indinavir. BMC Complement Altern Med. 2008 Aug 19;8:50. doi: 10.1186/1472-6882-8-50. PMID 18713456
- [Background] Barton DL, Soori GS, Bauer BA, Sloan JA, Johnson PA, Figueras C, Duane S, Mattar B, Liu H, Atherton PJ, Christensen B, Loprinzi CL. Pilot study of Panax quinquefolius (American ginseng) to improve cancer-related fatigue: a randomized, double-blind, dose-finding evaluation: NCCTG trial N03CA. Support Care Cancer. 2010 Feb;18(2):179-87. doi: 10.1007/s00520-009-0642-2. Epub 2009 May 6. PMID 19415341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from 2/13/13 through 10/19/15 from local HIV specialty clinics.
Pre-assignment Details: Participants who met study criteria returned for an enrollment visit for randomization. Study drugs (placebo or ginseng) were dispensed by the Investigational Pharmacy. Participants were instructed to take study drugs daily for 28 days. They returned 2 wks after finishing taking study drugs for a final visit. No wash out or run-in periods.
Groups:
- Placebo for American Ginseng 1000 mg/Day: 4-week of placebo for American ginseng 1000 mg/day every morning
  Placebo for American ginseng: Placebo for American ginseng 1000 mg/day and 3000 mg/day will be evaluated in the control arms for this study. Participants will be randomized to placebo for American ginseng 1000 or 3000 mg/day capsules taken daily for four weeks.
  Arms: Placebo for American ginseng 1000 mg/day, Placebo for American ginseng 3000 mg/day
- Placebo for American Ginseng 3000 mg/Day: 4-week of placebo for American ginseng 3000 mg/day every morning
  Placebo for American ginseng: Placebo for American ginseng 1000 mg/day and 3000 mg/day will be evaluated in the control arms for this study. Participants will be randomized to placebo for American ginseng 1000 or 3000 mg/day capsules taken daily for four weeks.
  Arms: Placebo for American ginseng 1000 mg/day, Placebo for American ginseng 3000 mg/day
Period: Overall Study
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Started | 32 | 17 | 31 | 16
Completed | 31 | 17 | 31 | 14
Not Completed | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants took the study product daily for 28 days. Participants returned 2 weeks after finishing taking the study product for a final evaluation. All participants completed questionnaires to quantify fatigue, were assessed for adverse events, and laboratory tests including inflammatory markers.
Groups:
- Total: Total of all reporting groups
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day | Total
Number analyzed (Participants) | 32 | 17 | 31 | 16 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (7.5) | 52.1 (9.5) | 53.7 (6.8) | 50.2 (4.83) | 52.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 13 | 9 | 44
  Male | 18 | 9 | 18 | 7 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 17 | 31 | 16 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Fatigue Severity Score (FSS)
Description: Change in FSS score from baseline to Week 4. The change in fatigue as measured by the FSS (Week 4 minus Baseline) using the Wilcoxon test. The FSS is a scale score ranging from 1 to 63 with higher scores indicative of more fatigue. A negative number indicates a decline in the FSS scale. Participants with FSS data at both times points were assessed.
Time Frame: From baseline to week 4 (28 days of study drugs)
Population: There was one missing scale from the ginseng 3000 arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 30 | 14
units on a scale | -24.7 (18.6) | -16.3 (18.6) | -16.9 (15) | -21.6 (16.0)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in the Brief Fatigue Inventory
Description: Questionnaire: Change in the Brief Fatigue Inventory (BFI) from baseline to week 4. We compared BFI scores from baseline to week 4 in the ginseng 1000 and 3000 mg arms with the combined placebo arms. We used the BFI Question that assess "Worst Fatigue" score: 0 to 90 scale. Higher scores means more fatigue; negative values mean less fatigue.The BFI was used to supplement the data obtained from the FSS.
Time Frame: Change in BFI scores from baseline to week 4 (28 days of study drugs)
Population: There was on missing questionnaire from the ginseng 3000 arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 30 | 14
units on a scale | -44.2 (34.3) | -26.5 (28.5) | -42.7 (32.4) | -37.9 (35.1)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.1329, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.1191, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Epworth Sleepiness Scale
Description: Questionnaire: Change in Epworth Sleepiness Scale (ESS) score from baseline to week 4. The ESS is scale ranges from 0 to 24; higher scores mean worse sleep disorder while a negative score indicates less sleep disorder. The ESS was used to supplement the data obtained from the FSS.
Time Frame: From baseline to week 4 (28 days of study drugs)
Population: There was one missing questionnaire from the ginseng 3000 arm
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 30 | 14
units on a scale | -5.74 (7.15) | -6.35 (4.43) | -6.97 (5.23) | -5.93 (3.17)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.7454, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.7391, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Patient Health Questionnaire 9
Description: Questionnaire: Change in Patient Health Questionnaire 9 (PHQ9) score from baseline to week 4. The scale for the PHQ9 score ranges from 0 to 27; higher scores mean worse depression; negative scores indicate less depression. We compared PHQ 9 scores from baseline to week 4 in the ginseng 1000 and 3000 mg arms with the combined placebo arms. The PHQ9 was used to supplement the data obtained from the FSS.
Time Frame: From baseline to week 4 (28 days of study drugs)
Population: There was one missed PHQ9 in the ginseng 3000 mg arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 30 | 14
units on a scale | -5.52 (4.76) | -5.59 (4.84) | -2.87 (4.20) | -3.86 (3.16)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.6818, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.0579, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Insomnia Severity Index
Description: Questionnaire: Change in Insomnia Severity Index (ISI) score from baseline to week 4. The ISI scale ranges from 0 to 28; higher scores mean worse insomnia while negative scores indicate less insomnia. The ISI was used to supplement the data obtained from the FSS.
Time Frame: From baseline to week 4 (28 days of study drugs)
Population: There was one missing ISI in the ginseng 3000 mg arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 30 | 14
units on a scale | -6.9 (6.07) | -5.47 (5.15) | -3.43 (5.49) | -3.57 (5.17)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Medical Outcomes Study HIV Health Survey
Description: Questionnaire: Change in Medical Outcomes Study (MOS) HIV Health Survey score from baseline to week 4. We evaluated the MOS Energy Fatigue scores; the MOS scale ranges from 0-100; higher scores mean more energy. The MOS was used to supplement the data obtained from the FSS.
Time Frame: From baseline to week 4 (28 days of study drugs)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 31 | 14
units on a scale | 22.4 (20.9) | 17.6 (19.5) | 24.0 (22.0) | 23.1 (21.3)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.7884, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.5532, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Changes in Clinical Global Impressions
Description: Questionnaire: Change in Clinical Global Impressions (CGI) scores from baseline to week 4. CGI is an instrument for making global assessments of worsening or improvement during interventional trials. The subject rates the change in the overall status since beginning the intervention (ranging from: very much improved, much improved, minimally improved, no change, and minimally worse). We assessed the number of participants who rated "very much improved".
Time Frame: From baseline to week 4 (28 days of study drugs)
Measure: Count of Participants; unit: Participants
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 31 | 14
Participants | 3 | 3 | 7 | 0
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.9885, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.2898, Wilcoxon (Mann-Whitney); 2 sides Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Inflammatory Markers
Description: Laboratory - Inflammatory Markers (IMs): Change in Interleukin (IL) -6 and soluble receptors of tumor necrosis factor (TNF) α 1 and 2 (sTNFR1 and sTNFR2) from baseline to week 4. Negative values indicate less change in inflammatory markers.
Time Frame: From baseline to week 4 (28 days of study drugs)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 31 | 14
pg/ml
  IL-6 | 0.22 (1.18) | 0.53 (1.99) | 0.079 (1.63) | 0.33 (1.33)
  sTNFR1 | 19.5 (135.5) | -15.5 (154.5) | 15.2 (170.5) | -6.24 (142)
  sTNFR2 | 183.5 (667.9) | 4.08 (580.5) | -207.7 (1156.1) | -201.7 (1156.1)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the IL-6 level changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the IL-6 level changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the sTNFR1 level changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the sTNFR1 level changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the sTNFR2 level changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the sTNFR2 level changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in CD4 Cell Count
Description: Laboratory: Change in absolute cluster of differentiation 4 (CD4) cell count from baseline to week 5. Negative values mean decline in CD4 cell count.
Time Frame: From baseline to week 5 (28 days of study drugs)
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 31 | 14
cells per cubic millimeter | 3.45 (111.5) | 56.6 (147.5) | -23.1 (148.4) | 34.4 (99.8)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 5 are significantly different between arms; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Plasma HIV RNA
Description: Laboratory: Change in plasma HIV RNA from baseline to week 4. A negative value means a drop in plasma HIV RNA.
Time Frame: From baseline to week 4 (28 days of study drugs)
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 31 | 14
copies/mL | 1.94 (6.19) | -0.06 (4.78) | 1.32 (7.02) | 0.0 (0.0)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in PROMIS Fatigue
Description: Questionnaire: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) fatigue score from baseline to week 4. Change in PROMIS fatigue score from baseline to Week 4. The change in fatigue as measured by the PROMIS fatigue (Week 4 minus Baseline) using the Wilcoxon test. The PROMIS fatigue is a scale with normalized mean of 50 and standard deviation (SD) of 10. Higher mean values mean more fatigue and negative values indicate less fatigue.
Time Frame: From baseline to week 4 (28 days of study drugs).
Population: There was one missed PROMIS fatigue questionnaire in the ginseng 3000 mg arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 31 | 17 | 30 | 14
units on a scale | -12.5 (11.8) | -11.1 (11.0) | -11.4 (10.9) | -9.49 (11.2)
Statistical Analysis 1: Comparison: American Ginseng 1000 mg/Day vs Placebo for American Ginseng 1000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo for American Ginseng 1000 mg/Day vs American Ginseng 3000 mg/Day vs Placebo for American Ginseng 3000 mg/Day; Testing whether the changes from baseline to week 4 are significantly different between arms; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney); 2 sided Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Number of Participants With Adverse Events in the Ginseng and Placebo Arms
Description: Adverse events (AEs) were assessed from baseline to wk 4 using the NIH Division of AIDS (DAIDS) Grading Toxicity Table, a well known tool used by NIH networks for assessing the severity of AEs in participants enrolled in clinical trials. Reporting the number of participants in each arm who experienced adverse events.
Time Frame: From baseline to week 4 (28 days of study drugs)
Measure: Count of Participants; unit: Participants
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
Number analyzed (Participants) | 32 | 17 | 31 | 16
Participants | 30 | 16 | 31 | 13

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: The NIH Division of AIDS Toxicity table was used to grade averse event severity for this clinical trial. Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Potentially Life Threatening), Grade 5 (Death). Some data was lost and is no longer available for 1 participant in the Ginseng 1000 mg/day arm, and 2 participants in the Placebo for the Ginseng 3000 mg/Day arm.
Arm/Group | American Ginseng 1000 mg/Day | Placebo for American Ginseng 1000 mg/Day | American Ginseng 3000 mg/Day | Placebo for American Ginseng 3000 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/17 | 0/31 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/32 | 2/17 | 4/31 | 2/16
Other Adverse Events (participants affected / at risk) | 30/32 | 16/17 | 31/31 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | American Ginseng 1000 mg/Day (N=32) | Placebo for American Ginseng 1000 mg/Day (N=17) | American Ginseng 3000 mg/Day (N=31) | Placebo for American Ginseng 3000 mg/Day (N=16)
Low ANC (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Low Absolute Neutrophil Count (ANC)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Bronchitis
Hip Replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Right Hip Replacement
Increased AST (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Increased Aspartate aminotransferase (AST)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hyperglycemia
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Cellulitis Right Finger
Pain Right Index Finger (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pain Right Index Finger
Kidney Stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Kidney Stone
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Abdominal Pain
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Ureterolithiasis
Right Flank Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Right Flank Pain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | American Ginseng 1000 mg/Day (N=32) | Placebo for American Ginseng 1000 mg/Day (N=17) | American Ginseng 3000 mg/Day (N=31) | Placebo for American Ginseng 3000 mg/Day (N=16)
anxiety (Psychiatric disorders) | 11 (11) | 9 (9) | 7 (7) | 5 (5) — Anxiety
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) — Cough
Decreased ANC (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 5 (5) | 3 (3) — Decreased ANC
Decreased Potassium (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) — Diarrhea
Diziness (Nervous system disorders) | 11 (12) | 7 (7) | 6 (6) | 5 (5) — Dizziness
Elevated ALT (Hepatobiliary disorders) | 7 (7) | 3 (3) | 6 (6) | 3 (3) — Elevated Alanine Aminotransferase (ALT)
Elevated AST (Hepatobiliary disorders) | 8 (8) | 4 (4) | 6 (6) | 4 (4) — Elevated AST
Elevated Alkaline Phosphatase (Hepatobiliary disorders) | 4 (4) | 4 (4) | 4 (4) | 1 (1) — Elevated Alkaline Phosphatase
Elevated Bilirubin (Hepatobiliary disorders) | 6 (6) | 1 (1) | 1 (1) | 2 (2) — Elevated Bilirubin
Elevated Creatinine (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) — Elevated Creatinine
Elevated Glucose (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (3) — Elevated Glucose
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) — Fatigue
Headache (Nervous system disorders) | 11 (13) | 9 (10) | 7 (14) | 5 (7) — Headache
Hypertension (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) — Hypertension
Insomnia (Nervous system disorders) | 11 (17) | 9 (9) | 7 (18) | 5 (5) — Insomnia
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 7 (9) | 5 (9) — Nausea
Nervousness (Nervous system disorders) | 9 (9) | 6 (6) | 5 (5) | 5 (5) — Nervousness
Upper Respiratory Infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 2 (2) — Upper Respiratory Infection
Hyperglycemia (Endocrine disorders) | 5 (5) | 4 (4) | 8 (8) | 4 (4) — Hyperglycemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No